CLINICAL TRIAL: NCT02285322
Title: Predictors of Blood Pressure Control and Associations With Cardiovascular Diseases in Individuals With High Blood Pressure: a CALIBER Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: Wellcome Trust (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Harry Hemingway, Professor of Epidemiology and Public Health, University College, London
Other Study IDs: 10_164R
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Stroke; Myocardial Infarction; Stable Angina Pectoris; Heart Failure
MeSH Terms: conditions — Stroke; Myocardial Infarction; Angina, Stable; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- BP control reached: Patients diagnosed with high blood pressure who lowered their blood pressure measurements during follow-up to <140/90mmHg if aged less than 60 years old, and <150/90mmHg for those of ≥60 years
- BP control not reached: Patients diagnosed with high blood pressure who did not lower their blood pressure measurement during follow-up (measurements were ≥140/90mmHg for individuals aged less than 60 years old, and ≥150/90mmHg for those of ≥60 years)

SUMMARY:
Current guidelines for the clinical management of hypertension in adults recommend to achieve and maintain blood pressure levels of <140/90 mmHg. However, it is uncertain what proportion of individuals identified with high blood pressure in primary care actually reach blood pressure control, what factors are associated with attainment of control and to what extent blood pressure control attainment is associated with cardiovascular diseases in a contemporary population of individuals diagnosed with high blood pressure.

The aim of this study is to investigate the extent to which patients achieve blood pressure control and associated risk factors, time to attainment of blood pressure control and whether this time is associated with an increased risk of CVD onset, all-cause and cardiovascular disease and end-stage renal disease.

DETAILED DESCRIPTION:
An increment of 20 mmHg of systolic blood pressure (or approximately equivalent 10 mmHg diastolic blood pressure) is associated with more than a two-fold increase in risk of fatal stroke, and with a two-fold increase in fatal ischemic heart diseases in individuals aged 40-69 years. The management and control of high blood pressure is therefore one of the most important components of primary and secondary strategies for prevention of cardiovascular mortality and morbidity. Current guidelines for the clinical management of hypertension in adults recommend to achieve and maintain blood pressure levels of <140/90 mmHg. However, it is uncertain what proportion of individuals identified with high blood pressure in primary care actually reach blood pressure control, what factors are associated with attainment of control and to what extent blood pressure control attainment is associated with cardiovascular diseases in a contemporary population of individuals diagnosed with high blood pressure. This is important for clinicians and policy decision makers in order to design and implement effective strategies for patient management.

The aim of this study is to investigate the extent to which patients achieve blood pressure control and associated risk factors, time to attainment of blood pressure control and whether this time is associated with an increased risk of CVD onset, all-cause and cardiovascular disease and end-stage renal disease.

The study will use data from the CALIBER data set of clinically collected electronic health record data from England.

This study is part of the CALIBER (Cardiovascular disease research using linked bespoke studies and electronic records) programme funded over 5 years from the National Institute for Health Research (NIHR) and Wellcome Trust. The central theme of the CALIBER research is linkage of the Myocardial Ischaemia National Audit Project (MINAP) with primary care (Clinical Practice Research Datalink - CPRD) and other resources. The overarching aim of CALIBER is to better understand the aetiology and prognosis of specific coronary phenotypes across a range of causal domains, particularly where electronic records provide a contribution beyond traditional studies. CALIBER has received both Ethics approval (ref 09/H0810/16) and ECC approval (ref ECC 2-06(b)/2009 CALIBER data set).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over
* Registered with a participating general practice during the study period
* Minimum one year of records prior to study entry meeting CPRD data quality
* Diagnosed with high blood pressure in the period January 1997 - March 2010

Exclusion Criteria:

* Patients without record of gender
* Patients with prior atherosclerotic disease, as recorded in primary care or hospitalisation data
* Patients with less than 6 months of follow-up since diagnosis of high blood pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in the CALIBER database who had high blood pressure (the Clinical Practice Research Datalink [CPRD]) and consenting to data linkage. High blood pressure was defined as the record of ≥3 systolic or diastolic high blood pressure readings within a one year period, or ≥2 systolic or diastolic high blood pressure readings within a 6 month period in CPRD. High blood pressure measurements were defined as in the eighth Joint National Committee (2014 JNC8) guidelines for patient management, that is ≥140/90mmHg for individuals aged less than 60 years old, and ≥150/90mmHg for those of ≥60 years.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
First presentation of cardiovascular disease | 10 years
  First recorded diagnosis of cardiovascular disease during follow-up: myocardial infarction, stroke (haemorrhagic or ischemic), heart failure, coronary revascularisation
All-cause mortality | 10 years
  Recorded death of any cause during follow-up
Cardiovascular mortality | 10 years
  Recorded death due to cardiovascular disease during follow-up
Risk factors for blood pressure control | 10 years
  Investigation of baseline factors associated with blood pressure control attainment during follow-up
Coronary revascularisation | 10 years
  First recorded percutaneous coronary intervention or coronary artery bypass graft (excluding interventions performed within 30 days before or after a diagnosis of myocardial infarction)

SECONDARY OUTCOMES:
First presentation of cardiovascular disease | 10 years
  First recorded diagnosis of cardiovascular disease during follow-up: stable angina pectoris and atrial fibrillation
End-stage renal disease | 10 years
  Recorded kidney disease resulting in dialysis or kidney transplantation during follow-up
Management of high blood pressure | 6 months after cohort entry
  Description of patient management in the 6 months after diagnosis of high blood pressure in terms of: blood pressure lowering medication start, timing and class; smoking cessation; dietary advice; physical activity; weight and total cholesterol decrease; and HDL-cholesterol increase

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, London, United Kingdom